CLINICAL TRIAL: NCT03235947
Title: Perioperative Disodium Fosfomycin in the Prophylaxis of Urinary Tract Infection in Kidney Transplant Recipients. Controlled Clinical Trial (PERIFOS Trial)
Brief Title: Perioperative Fosfomycin in the Prophylaxis of Urinary Tract Infection in Kidney Transplant Recipients
Acronym: PERIFOS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Laboratorios Senosiain, S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1649
Record Dates: First submitted 2017-06-06; First posted 2017-08-01 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Urinary Tract Infection; Asymptomatic Bacteriuria
Keywords: Renal transplant; Antimicrobian prophylaxis; Fosfomycin; Urinary tract infection; Asymptomatic bacteriuria
MeSH Terms: conditions — Urinary Tract Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Intervention Model Description: This is a randomized, parallel-group, controlled clinical trial conducted in a single center that will include renal transplant recipients over the age of 18 to assess the efficacy and safety of disodium fosfomycin in the perioperative period of renal transplantation. The intervention group will receive intravenous fosfomycin 4 g disodium three hours prior to: renal transplant surgery, removal of the urinary catheter and withdrawal of the ureteral catheter. The control group will receive placebo at the same time. Both groups will receive standard prophylaxis consisting of trimethoprim / sulfamethoxazole (160/800 mg) orally every 24 hours when the GFR is greater than 30 mL / min / 1.73m2.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fosfomycin disodium (Experimental): * Fosfomycin disodium 4 g intravenously: 3 hours before kidney transplant surgery, 3 hours before urinary catheter removal and 3 hours prior to ureteral catheter removal.
  * Trimethoprim / Sulfamethoxazole (160/800 mg) 1 tablet orally every 24 hours.
  Interventions: Drug: Fosfomycin disodium; Drug: Trimethoprim / Sulfamethoxazole
- Trimethoprim / Sulfamethoxazole (Active Comparator): * Trimethoprim / Sulfamethoxazole (160/800 mg) 1 tablet orally every 24 hours.
  * Intravenous placebo solution at the same time of application of fosfomycin disodium in the experimental arm.
  Interventions: Drug: Trimethoprim / Sulfamethoxazole; Drug: Intravenous placebo

INTERVENTIONS:
Drug: Fosfomycin disodium — Fosfomycin disodium 4 g intravenously dissolved in 100 mL of normal saline 0.9% three times in the perioperative period of renal transplant surgery.
  Arms: Fosfomycin disodium
Drug: Trimethoprim / Sulfamethoxazole — Trimethoprim / Sulfamethoxazole (160/800 mg) orally every 24 hours during the study follow-up (7 weeks)
Drug: Intravenous placebo — Normal saline 0.9% 100 mL intravenous administered three times in the perioperative period of the renal transplant, at the same times corresponding to disodium fosfomycin
  Arms: Trimethoprim / Sulfamethoxazole

SUMMARY:
A clinical controlled, randomized and double blind trial that included adult patients (≥18 years) receiving kidney transplantation (KT) at the INCMNSZ.

The intervention group will receive disodium fosfomycin 4 g intravenously in three moments: preoperative of transplant surgery, prior to removal of the urinary catheter and finally prior to removal of ureteral catheter. The control group will receive placebo in the same moments.

Both groups will receive prophylaxis standard for urinary tract infection (UTI), with trimethoprim/sulfamethoxazole 160/800 mg per day. This prophylaxis will be administered once the estimated glomerular filtration rate is greater than 30 mL/min/1.73m2.

The primary objective is to compare the average number of episodes of UTI´s and asymptomatic bacteriuria in both groups after 7 weeks of follow-up. The secondary objectives are to know the incidence of asymptomatic bacteriuria, the incidence of hospitalizations for IVU, the days of hospital stay, the pattern of bacterial resistance, the safety of disodium fosfomycin, and assessment of the function of the graft and rejection rate.

DETAILED DESCRIPTION:
In the context of development UTI in receptors of KT, some microbiological factors have raised great importance, mainly the antimicrobial drug resistance, which has been reported for TMP/SMX as high as 60 to 100%. Furthermore, it is also of increasing importance the recent isolation of multidrug-resistant bacteria, in particular ESBL-producing Escherichia coli and ampicillin-resistant Enterococcus. This phenomenon increases the rate of hospitalizations as well as the costs of hospital stay and antibiotic therapy. (1-3) In our institution, in receptors of KT the rate of TMP/SMX resistance is 89% and ESBL-production about 32% among E. coli recovered from urine. (4)

Because of the increase in the rate of TMP-SMX resistance, there is a lot of interest to use other antibiotics for the prevention of UTI among different populations. In this sense, fosfomycin is an agent with a unique mechanism of action that does not share with other families of known antibiotics, this characteristic provides advantages to use this antibiotic alone or, even, synergistically in combination with other antibiotics. Fosfomycin (FOS) is a wall antibiotic (pyruvyl-transferase inhibitor) that has shown a good bioavailability, especially in the urinary tract. It has shown a wide antibacterial spectrum, but the important target seems to be enteric bacilli particularly Escherichia coli (the most prevalent cause of UTI). FOS has also shown a very good activity against E. coli producer of Extended Spectrum Betalactamases.

Multiple clinical studies have shown FOS efficacy in the treatment of UTI's and especially in multiple-drug-resistant bacteria. (5) With regard to its use as a perioperative prophylaxis, in a systematic review with 8 trials, FOS proved to be effective to prevent health care-associated UTI's, however only one study showed no benefit. The oral dose regularly used is FOS 3 g, 3 hours before and 24 hours after the surgical procedure. (6)

Our hypothesis is that in the seven weeks after kidney transplantation, perioperative prophylaxis with FOS will show greater efficacy in comparison with standard prophylaxis (TMP/SMX). Considering that the mean number of UTI and BA episodes per patient in the first seven weeks is 0.8 episodes / patient, if we want to decrease it to 0.4 episodes per patient, using the means comparison formula will require 40 patients per arm per treatment, this considering a power of 80% and confidence intervals of 95%. The primary outcome will be to compare the mean number of episodes of urinary tract infection and asymptomatic bacteriuria per patient in each treatment arm. Secondary outcomes refer to the development of UTI-associated sepsis, pyelonephritis, recurrent UTI and asymptomatic bacteriuria. Safety outcomes included hematological and gastrointestinal side effects, the acute rejection rate, glomerular filtration rate, graft loss and patient death.

Patients eligible for a kidney transplant will be invited to participate in the study, prior to renal transplant surgery. They are given an informed consent, which is reviewed and approved by the ethics and research committees of our institution. The arms of the study are discussed in detail below. The study followed the Declaration of Helsinki recommendations and was approved by the Institutional Review Board (Ref: 1649). Randomization was conducted centrally by stratifying according to gender, with specific software (www.randomization.com). Patients were assigned to one of two parallel groups in a 1:1 ratio and in blocks of 4.

Subjects will be followed up for 7 weeks from renal transplant surgery. The outcome variables are defined as follows:

* Positive urine culture: The isolated germ will be defined depending on international standards. For enterobacteria and gram positive ≥100,000 colony-forming unit (CFU) / mL.
* Urinary tract infection: Positive urine culture plus presence of associated signs or symptoms.
* Significant Asymptomatic Bacteriuria: Will be identified from isolation ≥100,000 CFU/mL. In the case of women, the same insulation should be corroborated in a second urine culture sample.
* Asymptomatic Bacteriuria not significant: It will be identified from isolation of ≥1000 CFU/mL and will not be given antibiotic treatment.
* Hospitalization due to UTI: It will be defined as any UTI event that warrants hospitalization or that, having another reason for hospitalization, develop IVU that requires intravenous antimicrobial treatment.

The urine cultures will be taken from the first urine in the morning, obtaining the sample of medium jet with an approximate volume to collect of 25 to 50 mL. Urine samples were processed within the first hour after obtention.

The sample was inoculated in human blood agar and McConkey agar with a 1 microliter calibrated loop, and incubated at 35ºC, overnight. The report included the number of CFU. All clinical isolates were identified with the gram-negative and gram-positive identification cards by Vitek 2 (BioMérieux, Lyon, France) following the manufacturer´s instructions. AST-285 Vitek2 cards were used for gram-negative bacilli and the AST-591 Vitek2 card for gram-positive cocci (BioMérieux, Lyon, France); they were incubated and then interpreted by an expert in the system (version 7.01) and according to the Clinical & Laboratory Standards Institute (CLSI) M100-S24 (2014) guideline (20). Susceptibility to fosfomycin was determined by disk diffusion on cation-supplemented Müeller Hinton agar plates (CLSI, M07-A9); a bacterial suspension was inoculated in 0.5 mL Mc Farland, and a fosfomycin disk (200 micrograms [mcg]) supplemented with glucose-6-phosphate was used (50 mcg). Interpretation of inhibition halos in E. coli and Enterococcus faecalis isolates was based on CLSI M100-S24 (2014) criteria. The following were used as controls: E. coli ATCC 25922, E. coli ATCC 35218, Staphylococcus aureus ATCC 29213 and S. aureus ATCC 43300. Antimicrobial sensitivity to fosfomycin was determined with the microdilution broth method in E. coli, Klebsiella pneumoniae and Enterococcus spp. isolates. Müeller Hinton broth supplemented with glucose-6-phosphate (25 mcg/ml) was used, E. coli ATCC 25922, S. aureus ATCC 29213 and Pseudomonas aeruginosa ATCC 27853 were included as controls and results were interpreted according to the CLSI (M07-A10) and European Committee on Antimicrobial Susceptibility Testing (EUCAST) 2015 criteria (20,21).

Urine culture will be performed in the following situations: 1.- 48 hrs after the removal of the urinary catheter. 2.- Prior to removal of the ureteral catheter. 3.- At 4 weeks after renal transplantation. 4.- At 6 weeks after renal transplantation. 5.-In case of urinary storage symptoms suggestive of UTI or elevated creatinine (If the emergency department approach requires it). 6.- After antibiotic treatment of urinary tract infection or significant asymptomatic bacteriuria. In the case of women who have an episode of significant asymptomatic bacteriuria, this should be corroborated in two consecutive urine cultures.

Subjects will have the following follow-up visits: before ureteral catheter removal (first visit), 4 weeks of renal transplantation (second visit), 6 weeks (third visit) and one final visit at week 7.

Both follow-up visits and reports of urine cultures are recorded in the CRFs for each patient. In the follow-up consultations, adverse events will also be registered, if they are reported, are notified to the institutional committees and to the regulatory institutions of the health system of Mexico. An intermediate analysis will be carried out to determine both the effectiveness and safety of the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Patients transplanted in the Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran.

Exclusion Criteria:

* Allergy to Fosfomycin disodium or Trimethoprim / Sulfamethoxazole

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2016-09-07 (Actual); Primary Completion 2017-11-06 (Actual); Study Completion 2017-11-06 (Actual)

PRIMARY OUTCOMES:
To compare the efficacy of Fosfomycin-disodium/Trimethoprim-sulfamethoxazole with Placebo/Trimetoprim-sulfamexazol in the prophylaxis of urinary tract infection or significant asymptomatic bacteriuria among kidney transplantation recipients. | 7-weeks after transplantation
  The primary outcome in this clinical trial is the comparison of the mean number of episodes of urinary tract infection or significant asymptomatic bacteriuria, per patient in both arms of treatment among kidney transplantation recipients during the first seven weeks after surgery.

SECONDARY OUTCOMES:
The elapsed time period until the first urinary tract infection or asymptomatic bacteriuria developed | 7-weeks after transplantation
  Refers to the elapsed time period until the first urinary tract infection or asymptomatic bacteriuria developed during the first 7 weeks post-KT

OTHER OUTCOMES:
Incidence of urinary tract infection | 7-weeks after transplantation
  The number of patients that develope tract urinary infection in the first seven weeks after transplantation in each group, divided by the number of patients allocated in each group at randomization.
Incidence of asymptomatic bacteriuria | 7-weeks after transplantation
  The number of patients that develope asymptomatic bacteriuria in the first seven weeks after transplantation in each group, divided by the number of patients allocated in each group at randomization.
Incidence of bacteremia | 7-weeks after transplantation
  The number of patients that develope bacteremia in the first seven weeks after transplantation in each group, divided by the number of patients allocated in each group at randomization.
Incidence of hospitalization for urinary tract infection | 7-weeks after transplantation
  The number of patients that develope hospitalization for urinary tract infection in the first seven weeks after transplantation in each group, divided by the number of patients allocated in each group at randomization.
Incidence of Clostridium difficile infection | 7-weeks after transplantation
  The number of patients that develope Clostridium difficile infection in the first seven weeks after transplantation in each group, divided by the number of patients allocated in each group at randomization.
Incidence of multidrug resistant bacteria colonization | 7-weeks after transplantation
  The number of patients that develope multidrug resistant bacteria colonization infection in the first seven weeks after transplantation in each group, divided by the number of patients allocated in each group at randomization.
Incidence of acute rejection | 3-months after transplantation
  The number of patients that develope acute rejection in the first seven weeks after transplantation in each group, divided by the number of patients allocated in each group at randomization.

CONTACTS AND LOCATIONS:
Overall Officials: José Sifuentes-Osornio, MD, Principal Investigator — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Locations (1):
- Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided
The data would be available for future analysis for possible additional multicentered studies or metaanalysis.

REFERENCES:
- [Background] Linares L, Cervera C, Cofan F, Ricart MJ, Esforzado N, Torregrosa V, Oppenheimer F, Campistol JM, Marco F, Moreno A. Epidemiology and outcomes of multiple antibiotic-resistant bacterial infection in renal transplantation. Transplant Proc. 2007 Sep;39(7):2222-4. doi: 10.1016/j.transproceed.2007.06.061. PMID 17889144
- [Background] Kawecki D, Kwiatkowski A, Sawicka-Grzelak A, Durlik M, Paczek L, Chmura A, Mlynarczyk G, Rowinski W, Luczak M. Urinary tract infections in the early posttransplant period after kidney transplantation: etiologic agents and their susceptibility. Transplant Proc. 2011 Oct;43(8):2991-3. doi: 10.1016/j.transproceed.2011.09.002. PMID 21996207
- [Background] Senger SS, Arslan H, Azap OK, Timurkaynak F, Cagir U, Haberal M. Urinary tract infections in renal transplant recipients. Transplant Proc. 2007 May;39(4):1016-7. doi: 10.1016/j.transproceed.2007.02.060. PMID 17524879
- [Background] Figueroa-Sánchez G, Arreola-Guerra JM, Morales-Buenrostro LE. Time of presentation and antimicrobial resistance pattern of urinary tract infection in the early period after kidney transplantation. Rev Mex Traspl 2016; 5: 20-26.
- [Background] Falagas ME, Kastoris AC, Karageorgopoulos DE, Rafailidis PI. Fosfomycin for the treatment of infections caused by multidrug-resistant non-fermenting Gram-negative bacilli: a systematic review of microbiological, animal and clinical studies. Int J Antimicrob Agents. 2009 Aug;34(2):111-20. doi: 10.1016/j.ijantimicag.2009.03.009. Epub 2009 Apr 28. PMID 19403273
- [Background] Wagenlehner FM, Thomas PM, Naber KG. Fosfomycin trometamol (3,000 mg) in perioperative antibiotic prophylaxis of healthcare-associated infections after endourological interventions: a narrative review. Urol Int. 2014;92(2):125-30. doi: 10.1159/000355103. Epub 2013 Sep 13. PMID 24051657
- [Background] Clinical and Laboratory Standards Institute. Performance standards for antimicrobial susceptibility testing; twenty-fourth informational supplement. Document M100-S24. Wayne, PA: CLSI; 2014.
- [Background] The European Committee on Antimicrobial Susceptibility Testing. Breakpoint tables for interpretation of MICs and zone diameters. Version 6.0, 2016. http://www.eucast.org
- [Derived] Rosado-Canto R, Parra-Avila I, Tejeda-Maldonado J, Kauffman-Ortega C, Rodriguez-Covarrubias FT, Trujeque-Matos M, Cruz-Martinez R, Maravilla-Franco E, Criollo-Mora E, Arreola-Guerra JM, Morales-Buenrostro LE, Sifuentes-Osornio J. Perioperative fosfomycin disodium prophylaxis against urinary tract infection in renal transplant recipients: a randomized clinical trial. Nephrol Dial Transplant. 2020 Nov 1;35(11):1996-2003. doi: 10.1093/ndt/gfz261. PMID 31883327